CLINICAL TRIAL: NCT01870908
Title: Drug Use-result Survey to Assess the Safety and Efficacy of the Combination of Tacrolimus + Biological Agents in Daily Clinical Settings
Brief Title: Special Drug Use-Results Survey of Prograf Capsule in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PRGR03
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus; Biological Factors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tacrolimus + biological agents
  Interventions: Drug: tacrolimus; Drug: biological agents

INTERVENTIONS:
Drug: tacrolimus
  Other Names: prograf
Drug: biological agents

SUMMARY:
This study is to evaluate the safety and the effectiveness of treatment with tacrolimus and biological agents.

DETAILED DESCRIPTION:
The purpose of this study is to confirm the safety of 24 weeks-treatment with the combination of tacrolimus + biological agents, and to assess the efficacy using SDAI, CDAI, DAS28-CRP, MMP-3, MHAQ in patients with rheumatoid arthritis who have not achieved SDAI remission despite of using biological agents for over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis who have been treated with biological agents over 8 weeks but have not achieved SDAI remission (SDAI < 3.3)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who have been treated with biological agents
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Simplified disease activity index (SDAI) | Baseline and week-24

SECONDARY OUTCOMES:
Clinical disease activity index (CDAI) | Baseline, week-12 and week-24
Disease Activity Score 28 (DAS28) | Baseline, week-12 and week-24

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku